CLINICAL TRIAL: NCT04238806
Title: An Investigation of the Association Between Desflurane Inhalational Agent, Serum Brain Natriuretic Peptide (BNP) Levels and Clinical Outcomes During Coronary Artery Bypass Graft (CABG) Surgery
Brief Title: Desflurane,Brain Natriuretic Peptide and Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Collaborators: Trakya University Teaching and Research Hospital (Unknown)
Responsible Party: Principal Investigator, Ayse Baysal, Associate Professor, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2013.3/13
Record Dates: First submitted 2020-01-13; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Brain Natriuretic Peptide; Coronary Artery Bypass Graft Surgery; Cardiac Surgery; Cardiopulmonary Bypass; Desflurane; Outcome
MeSH Terms: interventions — Desflurane

STUDY DESIGN:
Intervention Model Description: In a prospective, randomized, double-blinded study, desflurane inhalational anesthesia was administered either continuously or intermittently (Group 1; n=60 versus Group 2; n=62).
Who Masked: Participant, Care Provider
Masking Description: The observers were blinded to the anesthetic protocol. Caregivers were not blinded, but they did not participate in data collection or data interpretation. Therefore, the study protocol is considered double-blinded, masked to observers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane Continuous (Active Comparator): In Group 1 of 60 patients, desflurane inhalational agent was administered continuously during coronary artery bypass graft surgery with cardiopulmonary bypass. Anesthesia induction was administered to all patients with intravenous midazolam at a dose of 0.2 mg/kg, fentanyl at a dose of 5 to 10 µg/kg and rocuronium bromide at a dose of 0.1 mg. For maintenance, in Group 1 patients, desflurane inhalational agent was administered at an end-tidal concentration of 1 to 4% during the whole surgical procedure and intravenous maintenance midazolam at a dose of 0.03 mg/kg and fentanyl at a dose of 1 to 2 µg/kg every half an hour. In Group 1 of patients, during the whole surgical procedure, attention to keep mean arterial pressure above 50 mmHg was provided.
  Interventions: Drug: Desflurane Inhalational agent
- Desflurane Intermittent (Active Comparator): In Group 2 of 60 patients, desflurane inhalational agent was administered intermittently during coronary artery bypass graft surgery with cardiopulmonary bypass. Anesthesia induction was administered to all patients with intravenous midazolam at a dose of 0.2 mg/kg, fentanyl at a dose of 5 to 10 µg/kg and rocuronium bromide at a dose of 0.1 mg/kg. For maintenance, in Group 2 patients, desflurane inhalational agent was administered at an end-tidal concentration of 1 to 4% before and after the cardiopulmonary bypass procedure as intermittently with the addition of intravenous maintenance midazolam at a dose of 0.03 mg/kg and fentanyl at a dose of 1 to 2 µg/kg every half an hour. In Group 2 of patients, during the whole surgical procedure, attention to keep mean arterial pressure above 50 mmHg was provided.
  Interventions: Drug: Desflurane Inhalational agent

INTERVENTIONS:
Drug: Desflurane Inhalational agent — Desflurane inhalational agent administration during the whole cardiac surgical operation with cardiopulmonary bypass versus administration of desflurane inhalational agent before and after cardiopulmonary bypass during the whole period of cardiac surgical operation.
  Other Names: Suprane

SUMMARY:
During coronary artery bypass grafting (CABG) operations with cardiopulmonary bypass (CPB), the use of desflurane continuously or intermittently may have effects on serum brain natriuretic peptide (BNP) levels. The aim is to investigate the association between desflurane, serum BNP values, and clinical outcomes during CABG operations. In a prospective, randomized, double-blinded study, desflurane inhalational anesthesia was administered either continuously or intermittently (Group 1; n=60 versus Group 2; n=62). The preoperative and postoperative BNP levels at 24, 48 and 72 hours after surgery were collected. Outcomes were recorded.

DETAILED DESCRIPTION:
Background: During coronary artery bypass grafting (CABG) operations with cardiopulmonary bypass (CPB), the use of desflurane continuously or intermittently may have effects on serum brain natriuretic peptide (BNP) levels.

Aim of the study: The aim is to investigate the association between desflurane, serum BNP values, and clinical outcomes during CABG operations.

Material and methods: In a prospective, randomized, double-blinded study, desflurane inhalational anesthesia was administered either continuously or intermittently (Group 1; n=60 versus Group 2; n=62). The preoperative and postoperative BNP levels at 24, 48 and 72 hours after surgery were collected. Outcomes were recorded. Randomization into two groups was performed using sealed envelopes. The sequentially numbered assignments of participants were concealed in these envelopes during the study. The patients enrolled in the study receive an allocation to a group after anesthesia induction by health care personnel after the opening of the envelope. The observers were blinded to the anesthetic protocol. Caregivers were not blinded, but they did not participate in data collection or data interpretation. Therefore, the study protocol is considered double-blinded, masked to observers. Inclusion criteria include; 18 to 75 years of age, body mass index of 25 to 31, ejection fraction≥50%. Exclusion criteria include; repeat cardiac surgery, emergent surgery, preoperative coagulation disorder, preoperative congestive heart failure, ejection fraction <49%, preoperative renal dysfunction (serum creatinine>1.3 mg/dL), dialysis, preoperative hepatic dysfunction (serum aspartate/alanine amino transferase>40 U/L), preoperative electrolyte imbalance, history of pancreatitis or current corticosteroid treatment.The primary endpoint was to determine preoperative and postoperative BNP values 24, 48 and 72 hours after surgery. The secondary endpoint was the relation between BNP values and clinical outcomes such as; 1-Aortic cross-clamp time, 2-Cardiopulmonary bypass time, 3-The use of inotropic support, 4-Intra-aortic balloon pump, 5-Duration of mechanical ventilation (>48 hours), 6-Development of pneumonia, 7-Perioperative myocardial infarction, 8-Cerebrovascular event (stroke or transient ischemic attack), seizure, 9-Atrial fibrillation and other rhythm disturbances, 10-Need for renal replacement therapy (RRT), 11-Reoperation secondary to bleeding, 12-Intensive care unit stay (>3 days), 13-Hospital stay and, 14-Thirty-day mortality.

Statistical analysis. The sample size was calculated according to the comparison of serum BNP values in a previous study and a sample size of 58 patients per group would be required with 80% power and the conventional 2-sided type 1 error of 5%. A multiple logistic regression analysis was performed to assess the predictive factors for weaning failure from mechanical ventilation, and the significance level was set at a p-value of less than 0.10 in the univariate model. To determine the best cut-off for preoperative BNP value to predict the development of prolonged mechanical ventilation, we calculated the area under the receiver operating characteristic curve.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen to seventy-five years of age,
* Body mass index values between twenty-five and thirty-one,
* Ejection fraction greater than or equal to 50%.

Exclusion Criteria:

* Repeat cardiac surgery,
* Emergent surgery,
* Preoperative coagulation disorder,
* Preoperative congestive heart failure,
* Ejection fraction less than 49%,
* Preoperative renal dysfunction (serum creatinine value of greater than 1.3 mg/dL),
* Dialysis,
* Preoperative hepatic dysfunction (serum aspartate/alanine amino transferase values of greater than 40 U/L),
* Preoperative electrolyte imbalance,
* History of pancreatitis,
* Current corticosteroid treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
Serum BNP values before the cardiac surgery | One day before cardiac surgery.
  Serum BNP values were collected from a blood sample of each patient one day before cardiac surgery
Serum BNP values after the cardiac surgery at 24 hours | After operation at 24 hours after cardiac surgery.
  Serum BNP values were collected from a blood sample of each patient after cardiac surgery
Serum BNP values after the cardiac surgery at 48 hours | After operation at 48 hours after cardiac surgery.
  Serum BNP values were collected from a blood sample of each patient after cardiac surgery
Serum BNP values after the cardiac surgery at 72 hours | After operation at 72 hours after cardiac surgery.
  Serum BNP values were collected from a blood sample of each patient after cardiac surgery
Serum BNP values before and after the cardiac surgery | After collection of the data and during statistical analysis
  The collected serum BNP values were compared with each other by repeated measure analysis

SECONDARY OUTCOMES:
Outcome aortic cross-clamp time | During operative time period of cardiac surgery
  A relation between serum BNP values and aortic cross-clamp time
Outcome cardiopulmonary bypass time | During operative time period of cardiac surgery
  A relation between serum BNP values and cardiopulmonary bypass time
Outcome use of inotropic support | During operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and use of inotropic support
Outcome use of Intra-aortic balloon pump | During operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and use of Intra-aortic balloon pump
Outcome duration of mechanical ventilation (>48 hours) | After operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and duration of mechanical ventilation (>48 hours)
Outcome development of pneumonia | After operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and development of pneumonia
Outcome parameters | During operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and perioperative myocardial infarction
Outcome cerebrovascular event or seizure | After operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and cerebrovascular event (stroke or transient ischemic attack) or seizure
Outcome atrial rhythm disturbances | After operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and atrial fibrillation and other atrial rhythm disturbances
Outcome ventricular rhythm disturbances | After operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and ventricular rhythm disturbances
Outcome renal replacement therapy | After operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and need for renal replacement therapy (RRT)
Outcome reoperation | After operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and reoperation secondary to bleeding
Outcome intensive care unit stay | After operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and intensive care unit stay (>3 days)
Outcome hospital stay | After operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and intensive care unit stay (>3 days)
Outcome thirty-day mortality | After operative time period of cardiac surgery and during intensive care unit stay
  A relation between serum BNP values and thirty-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Gonul Sagiroglu, MD, Study Director — Trakya University

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing plan includes sharing of the Study Protocol, Statistical Analysis Plan, and Statistical Analysis of the study with researchers upon request via e-mail.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The Study Protocol, the Clinical Study Report and the Statistical Analysis Plan are available after ClinicalTrials.gov registration.
Access Criteria: Accessible to all researchers

REFERENCES:
- [Result] De Hert SG, Cromheecke S, ten Broecke PW, Mertens E, De Blier IG, Stockman BA, Rodrigus IE, Van der Linden PJ. Effects of propofol, desflurane, and sevoflurane on recovery of myocardial function after coronary surgery in elderly high-risk patients. Anesthesiology. 2003 Aug;99(2):314-23. doi: 10.1097/00000542-200308000-00013. PMID 12883404
- [Result] Cuthbertson BH, Amiri AR, Croal BL, Rajagopalan S, Alozairi O, Brittenden J, Hillis GS. Utility of B-type natriuretic peptide in predicting perioperative cardiac events in patients undergoing major non-cardiac surgery. Br J Anaesth. 2007 Aug;99(2):170-6. doi: 10.1093/bja/aem158. Epub 2007 Jun 15. PMID 17573389
- [Result] Karthikeyan G, Moncur RA, Levine O, Heels-Ansdell D, Chan MT, Alonso-Coello P, Yusuf S, Sessler D, Villar JC, Berwanger O, McQueen M, Mathew A, Hill S, Gibson S, Berry C, Yeh HM, Devereaux PJ. Is a pre-operative brain natriuretic peptide or N-terminal pro-B-type natriuretic peptide measurement an independent predictor of adverse cardiovascular outcomes within 30 days of noncardiac surgery? A systematic review and meta-analysis of observational studies. J Am Coll Cardiol. 2009 Oct 20;54(17):1599-606. doi: 10.1016/j.jacc.2009.06.028. PMID 19833258
- [Result] Uhlig C, Bluth T, Schwarz K, Deckert S, Heinrich L, De Hert S, Landoni G, Serpa Neto A, Schultz MJ, Pelosi P, Schmitt J, Gama de Abreu M. Effects of Volatile Anesthetics on Mortality and Postoperative Pulmonary and Other Complications in Patients Undergoing Surgery: A Systematic Review and Meta-analysis. Anesthesiology. 2016 Jun;124(6):1230-45. doi: 10.1097/ALN.0000000000001120. PMID 27065094
- [Result] Yun KH, Jeong MH, Oh SK, Choi JH, Rhee SJ, Park EM, Yoo NJ, Kim NH, Ahn YK, Jeong JW. Preoperative plasma N-terminal pro-brain natriuretic peptide concentration and perioperative cardiovascular risk in elderly patients. Circ J. 2008 Feb;72(2):195-9. doi: 10.1253/circj.72.195. PMID 18219153
- [Result] Fox AA, Nascimben L, Body SC, Collard CD, Mitani AA, Liu KY, Muehlschlegel JD, Shernan SK, Marcantonio ER. Increased perioperative b-type natriuretic peptide associates with heart failure hospitalization or heart failure death after coronary artery bypass graft surgery. Anesthesiology. 2013 Aug;119(2):284-94. doi: 10.1097/ALN.0b013e318299969c. PMID 23695172
- [Result] Litton E, Ho KM. The use of pre-operative brain natriuretic peptides as a predictor of adverse outcomes after cardiac surgery: a systematic review and meta-analysis. Eur J Cardiothorac Surg. 2012 Mar;41(3):525-34. doi: 10.1093/ejcts/ezr007. Epub 2011 Oct 20. PMID 22345176
- [Result] Hutfless R, Kazanegra R, Madani M, Bhalla MA, Tulua-Tata A, Chen A, Clopton P, James C, Chiu A, Maisel AS. Utility of B-type natriuretic peptide in predicting postoperative complications and outcomes in patients undergoing heart surgery. J Am Coll Cardiol. 2004 May 19;43(10):1873-9. doi: 10.1016/j.jacc.2003.12.048. PMID 15145114
- [Result] Murad Junior JA, Nakazone MA, Machado Mde N, Godoy MF. Predictors of mortality in cardiac surgery: brain natriuretic peptide type B. Rev Bras Cir Cardiovasc. 2015 Mar-Apr;30(2):182-7. doi: 10.5935/1678-9741.20150008. PMID 26107449
- [Result] Lurati Buse GA, Koller MT, Burkhart C, Seeberger MD, Filipovic M. The predictive value of preoperative natriuretic peptide concentrations in adults undergoing surgery: a systematic review and meta-analysis. Anesth Analg. 2011 May;112(5):1019-33. doi: 10.1213/ANE.0b013e31820f286f. Epub 2011 Mar 3. PMID 21372274
- [Result] Cuthbertson BH, Croal BL, Rae D, Gibson PH, McNeilly JD, Jeffrey RR, Smith WC, Prescott GJ, Buchan KG, El-Shafei H, Gibson GA, Hillis GS. N-terminal pro-B-type natriuretic peptide levels and early outcome after cardiac surgery: a prospective cohort study. Br J Anaesth. 2009 Nov;103(5):647-53. doi: 10.1093/bja/aep234. Epub 2009 Aug 27. PMID 19713279